CLINICAL TRIAL: NCT03359759
Title: Evaluation of Efficiency in Cancerology of New Technologies as Telemedicine and Conected Objects (e-DomSanté)
Acronym: e-DomSanté
Status: Completed | Type: Observational
Sponsor: Institut Bergonié (Other)
Collaborators: Région Nouvelle Aquitaine (Unknown)
Responsible Party: Sponsor
Other Study IDs: IB2016-eDOMSANTE
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Results first posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: Telemedicine; Connected watches; Patient-Reported symptom monitoring; Secure Platform
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Conected objects — Every week, each patient report her symptoms and answer ten questions on the i-PAD. The connected watch reports the performance status (activtiy and time spent in bed or sitting), and the falls.
  If nurses or doctors detect any problem, they ask the patient for a telemedicine to try to help her. During the same time, nurses or doctors send a message on a secure plateform to the local team (nurse, General Practitioner, and pharmacists) and they reserve a place for an hospitalization if necessary.

SUMMARY:
Observational study about patients treated for a metastasis breast cancer who live far from their comprehensive cancer center and followed by telemedicine, connected watches and patient-reported symptom monitoring.

DETAILED DESCRIPTION:
The effectiveness of remote follow-up of cancer patients through weekly medicalquestionnaires filled in on their smartphone has been reported in international studies. Thesestudies demonstrated an improvement in quality of life (QoL) and survival of several months. Thee-DomSanté study proposes the combined use of innovative technological tools for theimprovement of patient care

This study was carried out with patients followed-up for metastatic breast cancer who lived far from their treatment center. They were offered, in addition to their usual follow-up, weekly medical questionnaires on an interactive tablet and aconnected watch that registered their falls, bedtime and their general activity. All this data arrive on a secure portal. In the event of an alert, telemedicine is organized by remote consultation with exchange on a secure platform, in parallel, between the center's carers and the treating physician, nurse, pharmacist or the Territorial Support Unit. The evaluation criteria used include telemedicine and patients' quality of life questionnaires as well as their satisfaction with care.

ELIGIBILITY:
Inclusion Criteria:

* Women more than 18 years old
* Treated for an advanced metastasis breast cancer
* Who live far from their comprehensive cancer center in the Landes department

Exclusion Criteria:

* Women who are not able to understand the study because of psychiatric disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for an advanced metastasis breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie QUENEL-TUEUX, MD, Principal Investigator — Institut Bergonié
Locations (1):
- Institut Bergonie, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Advanced Disease: Patients treated for an advanced metastasis breast cancer
Period: Overall Study
Arm/Group | Patients With Advanced Disease
Started | 15
Completed | 10
Not Completed | 5
Not completed — Death | 3
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Advanced Disease
Number analyzed (Participants) | 15
Age, Continuous [Mean (Full Range); unit: years] | 65 [36 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Region of Enrollment [Number; unit: participants]
  France | 15

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life of the Patients at 12 Months
Description: QoL assessed using the score of the FACT-B questionnaire. The FACT-B (Functional Assessment of Cancer Therapy - Breast) is a quality of life questionnaire used primarily with breast cancer patients. It is a validated tool used in both clinical and research settings.
  Total score range: 0-148 A higher score indicates better quality of life.
Time Frame: 12 months
Population: Patients alive, not lost to follow-up, and with a completed questionnaire
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Patients With Advanced Disease
Number analyzed (Participants) | 8
score on a scale | 59 [32 to 84]

2. Primary Outcome: Quality of Life of the Patients at 6 Months
Description: as for outcome 1
Time Frame: 6 months
Population: Patients alive, not lost to follow-up, and with a completed questionnaire
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Patients With Advanced Disease
Number analyzed (Participants) | 11
score on a scale | 58 [33 to 77]

ADVERSE EVENTS:
Time Frame: 12 months. Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Description: Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Arm/Group | Patients With Advanced Disease
All-Cause Mortality (participants affected / at risk) | 3/15
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes